CLINICAL TRIAL: NCT05281991
Title: Agreement Between Laterality of Tsui Test and Laterality of Color Flow Doppler Signals During Labor Epidural Analgesia: a Prospective Observational Study
Brief Title: Agreement Between Laterality of Tsui Test and Laterality of Color Flow Doppler Signals During Labor Epidural Analgesia
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 22-01
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Labor Pain
Keywords: epidural catheter; epidural analgesia; labor epidural; ultrasound; Doppler; Tsui test
MeSH Terms: conditions — Labor Pain | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who had an epidural placed for labour: Patients who had an epidural placed for labour may take part. Study procedures will take place after delivery and prior to removal of the epidural catheter.
  Interventions: Device: Doppler ultrasonography; Device: Tsui test

INTERVENTIONS:
Device: Doppler ultrasonography — color flow Doppler ultrasonography
Device: Tsui test — The stimulator is set at frequency of 1Hz with 0.2 msec pulse width and the current output ranging from 0 to 20 mA. The current output will be carefully increased from zero until motor activity is detected up to a maximum of 20 mA.

SUMMARY:
Epidural analgesia for relief of labor pain is a very common, safe and reliable technique that requires placement of a catheter in the epidural space. About 5% of labor epidural catheters may need to be re-sited due to failure of analgesia. This is often caused by malposition of the epidural catheter. Many factors may influence the position of the tip of the epidural catheter and the resulting spread of local anesthetic solution within the epidural space and consequently the quality of labor pain management. The electrical stimulation of the epidural catheter, commonly known as Tsui test, can reliably confirm its positioning within the epidural space if this stimulus produces a muscular twitch under a certain current amplitude threshold. This muscular response is unilateral in 90% of the cases, not having any relationship between unilaterality and unsatisfactory catheter performance. It is unknown if this unilateral response has any correlation with the actual position of the catheter tip in terms of right or left side of the epidural space. Furthermore, the Tsui test does not give any information on the spread of anesthetic solution into the epidural space. Recent investigation shows that color flow doppler ultrasound during fluid injection through the epidural catheter may be helpful in determining the laterality of the tip of the epidural catheter; furthermore it may be able to inform about the spread the anesthetic solution, which is a limitation of the Tsui test. The investigators will perform an observational study to investigate the response patterns of Tsui test and Color flow Doppler ultrasound in the obstetric population. Women who have delivered under epidural analgesia will be approached for the study before the epidural catheter is removed. The investigators aim to characterize the laterality and current thresholds of Tsui test response and the laterality of the lumbar epidural catheter tip by color doppler ultrasound. The investigators hope to describe the findings and to correlate them with other clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have delivered vaginally under epidural anesthesia

Exclusion Criteria:

* Patients who refuse, are unable to give or have withdrawn consent
* Patients unable to communicate fluently in English.
* Patients who experience fetal or maternal complications during delivery.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who have delivered vaginally under epidural analgesia will be approached for the study before the epidural catheter is removed.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Tsui test motor response: questionnaire | 5 minutes
  Tsui test motor response will be recorded as either: left, right or bilateral
Colour flow Doppler ultrasound assessment: questionnaire | 5 minutes
  Colour flow Doppler ultrasound assessment will be recorded as either: left, right or bilateral

SECONDARY OUTCOMES:
Tsui test current threshold amplitude | 5 minutes
  Epidural catheter stimulation will be performed in all patients with a 0.2 msec pulse width and 1 Hz frequency. The current will be increased from 0 mA until a motor response is observed or until the maximum current of 20 mA is reached.
Tsui test motor response dermatome: abdomen, thigh, leg, feet | 5 minutes
  The muscle group involved in the response will be documented as: abdomen, thigh, leg, feet.
  Whether right, left or bilateral will also be recorded.
Location of epidural catheter tip flow as detected by Doppler | 5 minutes
  Location (interspace) of epidural catheter tip flow as detected by Doppler.
Need for catheter mobilization: questionnaire | 12 hours
  The need for catheter mobilization, including replacement (at any time after it is placed) will be documented as yes or no.
Presence of asymmetric block: questionnaire | 12 hours
  The presence of asymmetric block (>=2 segments difference) will be documented as yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada